CLINICAL TRIAL: NCT05220969
Title: Total Genotype Score, Growth, Maturation and Loading Exposure as Risk Factors for Injury in Elite Male Youth Football
Status: Completed | Type: Observational
Sponsor: St Mary's University College (Other)
Collaborators: Fulham Football Club (Unknown)
Responsible Party: Sponsor
Other Study IDs: SMEC_2019-20_003
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Fractures in Children; Apophysitis; Muscle Strain; Ligament Injury; Tendon Injuries; Genetic Predisposition
MeSH Terms: conditions — Sprains and Strains; Tendon Injuries; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite male youth footballers: Elite male youth footballers at an English championship / premier league football club
  Interventions: Genetic: Total Genotype Risk Score

INTERVENTIONS:
Genetic: Total Genotype Risk Score — A total genotype risk score has been generated based on the results of previously observed genetic association studies

SUMMARY:
A total genotype risk score was generated based on the findings of previous research for non-contact injury, non-contact muscle injury, tendon injury, ligament injury, fracture injury and apophysitis injury. This score was then compared with the incidence of injury between those with high, medium and low risk scores for each injury. The influence of different rates of growth, stages of physical maturation and loading exposure were then also included in the risk model to see if any interaction effects could be observed between genetic risk score and susceptibility to injury in different categories of growth, maturation and loading exposure.

ELIGIBILITY:
Inclusion Criteria:

* Elite male football players

Exclusion Criteria:

* Female
* non-elite

Ages: 12 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Elite male football players aged 12-40
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Fracture Injury Risk | 8 Years
  Did the risk of fracture differ between total genotype risk score categories? was this affected by maturation?
Non-Contact Injury Risk | 8 Years
  Did the risk of non-contact injury differ between total genotype risk score categories? was this affected by maturation, and loading?
Non-Contact Muscle Injury Risk | 8 Years
  Did the risk of non-contact muscle injury differ between total genotype risk score categories? was this affected by maturation, and loading?
Tendon Injury Risk | 8 Years
  Did the risk of tendon injury differ between total genotype risk score categories? was this affected by maturation, and loading?
Ligament Injury Risk | 8 Years
  Did the risk of ligament injury differ between total genotype risk score categories? was this affected by maturation?
Apophysitis Injury Risk | 8 Years
  Did the risk of ligament injury differ between total genotype risk score categories? was this affected by maturation?

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Fulham Football Club, London, New Malden
  - St Mary's University, Twickenham, London, Twickenham